CLINICAL TRIAL: NCT01614262
Title: Examining the Role of Continuous Glucose Monitoring (CGM) in Non-Insulin Treated Type 2 Diabetes
Brief Title: Examining The Role of CGM in T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Medtronic (Industry); Atlanta Diabetes Associates (Other); UNC Coordinating Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-0899
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2015-07

CONDITIONS: DIABETES MELLITUS, NONINSULIN-DEPENDENT, 2 (Disorder)
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Glucose Monitoring (Experimental): The Continuous Glucose Monitoring (CGM) arm will receive care based upon results from there CGM data; treatment decisions are based on algorithm and CGM data
  Interventions: Other: Continuous Glucose Monitoring with treatment algorithm
- Self Monitoring Blood Glucose (Active Comparator): Subjects in the Self Monitoring Blood Glucose group will have treatment decisions based on self monitored blood glucose values and not CGM values, per current standard of care.
  Interventions: Other: Continuous Glucose Monitoring with treatment algorithm

INTERVENTIONS:
Other: Continuous Glucose Monitoring with treatment algorithm — those subjects randomized to Continuous Glucose Monitoring results will be placed in CareLink iPro Clinical Management system, the experimental treatment guideline/algorithm has been programmed into the system. Providers will make treatment decisions based off of results of CGM.

SUMMARY:
Continuous glucose monitoring (CGM) technology has advanced the treatment of people with diabetes, however to date this technology had been primarily limited to use in patients treated with insulin. CGM is a powerful tool that has the potential to enhance the care of patients treated with agents other than insulin; however this has not been tested. The purpose of this study is to determine whether improved glycemic control can be achieved through the use of intensive, periodic CGM monitoring in patients with T2DM treated with oral anti-hyperglycemic drugs (OADs). The data gathered from this pilot study will be utilized to determine if a larger, clinical effectiveness study to assess use of CGM to improve clinical outcomes in patients with T2DM treated with OADs is warranted.

DETAILED DESCRIPTION:
The study will enroll and follow 90 participants for 187 days at two sites. Participants will be randomized (1:1 allocation ratio) to the CGM based intervention (Group 1) or the Self-Monitoring Blood Glucose (SMBG) based intervention (Group 2). Group 1 will receive care based upon the results of their CGM data while group 2 will receive care based upon traditional SMBG values. The clinical management algorithm will be utilized to guide the care of all subjects. All study participants will receive the iPro 2 devices (Medtronic Minimed, Northridge, CA 91325) to collect glucose measurements during five 1 week periods beginning on Day 0, Day 45, Day 90, Day 135 and Day 180. Laboratory measures of glucose control (HbA1c and FPG) and quality of life outcomes will be evaluated at Day 0, Day 90 and Day 187.

The iPro2 device is FDA approved for sale in the US and is a commercial product. The iPro2 digital recorder is intended to continuously record interstitial glucose levels in persons with diabetes mellitus. The iPro 2 is intended to be worn for intermittent periods to uncover glycemic variability and patterns. The data obtained can then be used to maximum treatment strategies to improve patient outcomes. The advantage to the iPro 2 is that it is blinded and will not be influenced by the patient.

The Enlite sensor, is an investigational device, is a 6 day sensor. The subjects in this study will wear the Enlite sensor for a 6 day monitoring period. The Enlite sensor is CE-marked and available for sale in over 50 countries and is currently seeking FDA approval.

CareLink iPro Clinical Therapy Management Software is part of the iPro2 CGM system. The Carelink iPro Clinical Software is intended to support clinical trials. This internet based software allows data to be viewed and easily evaluated by physicians. A PC links to Carelink iPro Clinical via the Internet and allows the user to upload data from Medtronic Diabetes iPro2 devices. Because the algorithm proposed in this protocol has been programed into the Software, this is an (IDE-exempt) investigational device.

Adult individuals 18-70 years of age, diagnosed with T2DM who are currently being treated in the Principal Investigators or referring physicians practice with a HbA1c between 7.5-9.0%.

ELIGIBILITY:
Inclusion Criteria:

* A subject is eligible for the study if all of the following criteria are met:

  1. Provide written informed consent prior to enrollment
  2. Is male or female between 18-70 years old
  3. Has been treated by the Principal Investigator or referring physician in the same practice.
  4. Has Type 2 Diabetes Mellitus for greater than 12 months on 1-3 antihyperglycemic medications, on a stable dose for 90 days prior to screening.
  5. Has a HbA1c between 7.5-9.0% in the 90 days prior to screening.
  6. Currently performs self-monitoring blood glucose checks at least 3 times per week.
  7. Ability to adhere to protocol requirements.

Exclusion Criteria:

* 1. Has Type 1 Diabetes or Gestational Diabetes

  2.Is pregnant or planning to become pregnant during the course of the study.

  3.Current use of any insulin or history of insulin use in the last 6 months.

  4.An acute coronary or cerebrovascular event in the previous 3 months.

  5.Any planned surgery during the course of the study.

  6.Current continuous renal replacement therapy.

  7.BMI ≥ 45 kg/m^2

  8.Current oral or injectable steroid use.

  9.Any previous history Continuous Glucose Monitoring use by any device or manufacturer.

  10.Has a serious or unstable medical or psychological condition which, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
change in glycosylated hemoglobin using intensive periodic CGM monitoring vs traditional monitoring | baseline and day 187

SECONDARY OUTCOMES:
change in fasting plasma glucose between two groups | baseline and day 187
comparison of change of the area under the curve for CGM results for both treatment arms | baseline and day 187
quality of life data evaluation | baseline and day 187
  Provide preliminary data on the effect of CGM monitoring on subjects' quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: John B Buse, MD, PhD, Principal Investigator — University of North Carolina
Locations (2):
- United States (2):
  - Atlanta Diabetes Assoicates, Atlanta, Georgia
  - University of North Carolina, Chapel Hill, North Carolina